CLINICAL TRIAL: NCT02470208
Title: A Prospective Observational Trial to Evaluate Hematopoietic Stem Cell Transplantation CMV Reactivation Events - Assessed by a CMV-Specific T-SPOT Assay: The REACT Study
Brief Title: Observational Trial to Evaluate Hematopoietic Stem Cell Transplantation CMV Reactivation
Acronym: REACT
Status: Completed | Type: Observational
Sponsor: Oxford Immunotec (Industry)
Responsible Party: Sponsor
Other Study IDs: US OI 125
Record Dates: First submitted 2015-06-03; First posted 2015-06-12 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2016-06

CONDITIONS: Infection
Keywords: Cytomegalovirus reactivation in stem cell transplant
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the ability of the T-SPOT.CMV assay to determine immune competence against CMV infection in stem cell transplantation.

To determine the utility of the T-SPOT.CMV assay used before transplantation to determine immune competence against subsequent CMV reactivation and to determine the utility of the T-SPOT.CMV assay used after transplantation to determine immune competence against subsequent CMV reactivation.

DETAILED DESCRIPTION:
In this prospective, non-randomized, observer-blind observational study, up to 200 patients who meet the study's eligibility criteria will be enrolled at up to 20 study centers. Enrollment will be actively managed by the sponsor.

Blood samples will be collected up to 14 days before transplantation, and then at 2-week intervals for the 6 months after the transplant procedure.

Study duration: 15 months: 9 months to enroll all patients, with 6 months (182 days) of participation for each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patients who will undergo one of the following types of allogeneic transplantation: matched related donor, matched or mismatched unrelated donor, haploidentical, or cord blood.
3. Patients must be seropositive for CMV prior to transplantation, regardless of donor seropositivity.
4. Institutional Review Board (IRB)-approved written Informed Consent and privacy agreement per national regulation (e.g., Health Insurance Portability and Accountability Act [HIPAA] for sites in the USA) must be obtained from the patient or the patient's legally authorized representative prior to any study-specific procedures.
5. Patients must be considered suitable for the study by the Investigator.

Exclusion Criteria:

* 1. Patients with a known active CMV reactivation within 1 month prior to enrollment or during the study's pre-transplant screening period.

  2. Patients who have received any antiviral therapy active against CMV other than acyclovir and valacyclovir (i.e., foscarnet, ganciclovir, valganciclovir, or cidofovir) during the month prior to enrollment.

  3. Patients who have previously received or are planning to receive a CMV vaccine.

  4. Patients who are known to be hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) positive.

  5. Patients who are known to have a clinically significant medical or psychiatric condition considered a high risk for participation in an investigational study.

  6. Patients who are participating in or plan to participate in CMV-related drug or vaccine studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in this study will be men or women aged 18 years or older with positive CMV serostatus (R+) who are candidates for allogeneic HSCT.
  The patients enrolled are intended to be representative of those who would be anticipated to have T SPOT.CMV testing when it is used in routine clinical practice. Enrollment will be actively managed by the sponsor.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-06; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of the T SPOT.CMV assay to determine immune competence against CMV infection in stem cell transplantation. | up to day 182
  change in T-SPOT counts from baseline to 182 days post transplant

SECONDARY OUTCOMES:
To determine the utility of the T SPOT.CMV assay used before transplantation to determine immune competence against subsequent CMV reactivation. | up to day 182
  change in T-SPOT counts from baseline to 182 days post transplant
To determine the utility of the T SPOT.CMV assay used after transplantation to determine immune competence against subsequent CMV reactivation. | up to day 182

CONTACTS AND LOCATIONS:
Overall Officials: Roy F Chemaly, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (12):
- United States (10):
  - City of Hope, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - The University of Chicago Medicine, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Wayne State University - School of Medicine, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- University Health Network, Toronto, Ontario, Canada
- Karolinska Univeristy Hostpital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided